CLINICAL TRIAL: NCT01770379
Title: A Phase III Randomized, Double-blind, Placebo-controlled Multicenter Study of Subcutaneous Secukinumab in Prefilled Syringes to Demonstrate the Efficacy at 24 Weeks and to Assess the Long Term Efficacy, Safety, Tolerability and Usability up to 5 Years in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Anti-TNFα Agents
Brief Title: Secukinumab Efficacy and Safety Study in Patients With Rheumatoid Arthritis and Inadequate Response to Anti-TNFα Agents.
Acronym: REASSURE2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457F2311; 2011-006058-94 (EudraCT Number)
Record Dates: First submitted 2012-10-16; First posted 2013-01-17 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, RA, IL-17 blocker, subcutaneous, self-injection, AIN457, AIN457F, secukinumab, anti-TNFα, pre-filled syringe
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Secukinumab 75 mg (Experimental): Secukinumab 75 mg s.c.
  Interventions: Biological: Secukinumab (AIN457)
- Secukinumab 150 mg (Experimental): Secukinumab 150 mg s.c.
  Interventions: Biological: Secukinumab (AIN457)
- Placebo (Placebo Comparator): Placebo patients will be re-randomized 1:1 to secukinumab 75 or 150mg s.c. (non-responders at Week 16 will be re-assigned to new treatment at Week 16; responders at Week 16 will be re-assigned to new treatment at Week 24)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab (AIN457) — Secukinumab is a human monoclonal antibody. Monoclonal antibodies are proteins that recognize and bind to unique proteins that your body produces. Secukinumab binds and reduces the activity of a cytokine (a "messenger" protein in the body) called Interleukin 17 (IL-17)
  Other Names: AIN457
  Arms: Secukinumab 150 mg; Secukinumab 75 mg
Biological: Placebo
  Arms: Placebo

SUMMARY:
This study will provide efficacy and safety data of the secukinumab pre-filled syringe (PFS) for subcutaneous self-administration in patients with active rheumatoid arthritis who are intolerant to or have had an inadequate response to anti-TNF-α agents.

ELIGIBILITY:
Inclusion Criteria: • Presence of Rheumatoid Arthritis classified by ACR 2010 revised criteria for at least 3 months •Disease activity defined by ≥6 tender joints out of 68 and ≥ 6 swollen joints out of 66 at baseline and with: Either Anti-CCP antibodies positive OR Rheumatoid Factor positive AND WITH Either hsCRP ≥ 10 mg/L OR ESR ≥28 mm/1st hr •Intake of at least one anti-TNF-α agent such as etanercept, adalimumab, infliximab, certolizumab or golimumab for at least 3 months before entering the study and to have experienced an inadequate response to treatment or to have been intolerant to at least one administration Exclusion Criteria:

* Current RA functional status class IV according to the ACR 1991 revised criteria •Previous use of secukinumab or other biologic drug directly targeting IL-17 or IL-17 receptor and/or any history of hypersensitivity to secukinumab or its excipient or to drugs of similar chemical classes. Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (71):
- United States (23):
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pembroke Pines, Florida
  - Novartis Investigative Site, Zephyrhills, Florida
  - Novartis Investigative Site, Cumberland, Maryland
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Tupelo, Mississippi
  - Novartis Investigative Site, Lees Summit, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Zanesville, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Benbrook, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Mesquite, Texas
- Argentina (3):
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Brazil (4):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, São Paulo, São Paulo
- Colombia (2):
  - Novartis Investigative Site, Cali, Colombia
  - Novartis Investigative Site, Bogotá
- Czechia (2):
  - Novartis Investigative Site, Uherské Hradiště, Czech Republic
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Santo Domingo, Republica Dominicana, Dominican Republic
- Germany (6):
  - Novartis Investigative Site, Hanover, Germany
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Pirna
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Heraklion, GR
  - Novartis Investigative Site, Athens
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- India (4):
  - Novartis Investigative Site, Secunderabad, Andhra Pradesh
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
- Italy (5):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Bologna
- Japan (13):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Takasaki, Gunma
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Miyagi-gun, Miyagi
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Setouchi, Okayama-ken
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Toyama, Toyama
- Novartis Investigative Site, Panama City, Provincia de Panamá, Panama
- Novartis Investigative Site, Lisbon, Portugal, Portugal
- Novartis Investigative Site, Panorama, Western Cape, South Africa
- Novartis Investigative Site, Seoul, Korea, South Korea

REFERENCES:
- [Derived] Huang Y, Fan Y, Liu Y, Xie W, Zhang Z. Efficacy and safety of secukinumab in active rheumatoid arthritis with an inadequate response to tumor necrosis factor inhibitors: a meta-analysis of phase III randomized controlled trials. Clin Rheumatol. 2019 Oct;38(10):2765-2776. doi: 10.1007/s10067-019-04595-1. Epub 2019 May 14. PMID 31087226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients received AIN457 75 mg, AIN457 150 mg or placebo as subcutaneous (s.c.) loading dose once weekly at baseline (BSL), Weeks 1, 2, 3 and 4, followed by monthly maintenance starting at Week 4.
Pre-assignment Details: At Wk 16, patients were classified as responders or non-responders. Placebo patients who were non responders were rerandomized at Wk 16 to AIN457 75 mg or AIN457 150 mg (1:1). Patients on placebo who were responders continued to receive placebo until Wk 24, these patients were re-randomized to receive AIN457 75 mg or AIN457 150 mg (1:1).
Groups:
- AIN457 75 mg: 75 mg secukinumab: Patients on secukinumab 75 mg continued to receive secukinumab 75 mg via PFS every 4 weeks regardless of responder status.
- AIN457 150mg: 150 mg secukinumab: Patients on secukinumab 150 mg continued to receive secukinumab 150 mg via PFS every 4 weeks regardless of responder status.
- Placebo: At Wk 16, patients were classified: responders or non-responders. Placebo patients who were non responders were rerandomized at Wk 16 to AIN457 75 mg or AIN457 150 mg (1:1). Patients on placebo who were responders continued to receive placebo until Wk 24, these patients were re-randomized to receive AIN457 75 mg or AIN457 150 mg (1:1)
Period: Overall Study
Arm/Group | AIN457 75 mg | AIN457 150mg | Placebo
Started | 80 | 81 | 81
Completed | 41 | 37 | 39
Not Completed | 39 | 44 | 42
Not completed — Technical issues | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 10 | 7
Not completed — study terminated by sponsor | 22 | 23 | 22
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Lack of Efficacy | 8 | 6 | 6
Not completed — Adverse Event | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 75 mg | AIN457 150mg | Placebo | Total
Number analyzed (Participants) | 80 | 81 | 81 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 70 | 62 | 69 | 201
  >=65 years | 10 | 19 | 12 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 67 | 65 | 202
  Male | 10 | 14 | 16 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an American College of Rheumatology Response 20 (ACR20).
Description: ACR20 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 20% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR).
  The ACR20 response results at week 24 used non-responder imputation.
Time Frame: Week 24
Population: Full analysis set (FAS): The FAS was comprised of all patients from the randomized set to whom study treatment had been assigned.
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 75 mg | AIN457 150mg | Placebo
Number analyzed (Participants) | 80 | 81 | 81
percentage of participants | 37.5 | 38.3 | 27.2
Statistical Analysis 1: Comparison: AIN457 75 mg vs Placebo; Test type: Superiority or Other; p = 0.2001, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.79 to 3.03]
Statistical Analysis 2: Comparison: AIN457 150mg vs Placebo; Test type: Superiority or Other; p = 0.1574, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.83 to 3.15]

2. Secondary Outcome: Change From Baseline in Disease Activity Score Utilizing CRP (DAS28-CRP)
Description: The DAS28 is a measure of disease activity in RA based on Swollen and Tender Joint Counts (out of a total of 28), hsCRP and the Patient's Global Assessment of Disease Activity. A DAS28 score greater than 5.1 implies active disease, equal to or less than 3.2 low disease activity, and less than 2.6 remission. A negative change from baseline indicates improvement.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AIN457 75 mg | AIN457 150mg | Placebo
Number analyzed (Participants) | 80 | 81 | 81
Units on a scale | -1.56 (0.149) | -1.61 (0.148) | -1.01 (0.176)

3. Secondary Outcome: Change From Baseline in Stanford Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in 8 categories of functioning including dressing, rising, eating, walking, hygiene, reach, grip and usual activities. The stem of each item asks 'Over the past week, "are you able to..." perform a particular task'. Each item is scored on a 4 point scale from 0 - 3, representing normal, no difficulty (0), some difficulty (1), much difficulty (2) and unable to do (3). The disability index score is calculated as the mean of the available category scores, ranging from 0 to 3. A negative change from baseline indicates improvement.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- AIN457 150 mg: 150 mg secukinumab: Patients on secukinumab 150 mg continued to receive secukinumab 150 mg via PFS every 4 weeks regardless of responder status.
Arm/Group | AIN457 75 mg | AIN457 150 mg | Placebo
Number analyzed (Participants) | 80 | 81 | 81
units on a scale | -0.42 (0.068) | -0.39 (0.068) | -0.13 (0.078)

4. Secondary Outcome: Percentage of Participants Achieving ACR50
Description: ACR50 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 50% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR).
  The ACR50 response results at week 24 used non-responder imputation.
Time Frame: Week 24
Population: Full analysis set: the full analysis set was comprised of all randomized participants (excluding mis-randomized participants) who were assigned to study treatment
Measure: Number; unit: Percentage of patients
Arm/Group | AIN457 75 mg | AIN457 150mg | Placebo
Number analyzed (Participants) | 80 | 81 | 81
Percentage of patients | 17.5 | 18.5 | 13.6

ADVERSE EVENTS:
Groups:
- Any AIN457 75 mg: 75 mg secukinumab: Patients on secukinumab 75 mg continued to receive secukinumab 75 mg via PFS every 4 weeks regardless of responder status.
- Any AIN457 150 mg: 150 mg secukinumab: Patients on secukinumab 150 mg continued to receive secukinumab 150 mg via PFS every 4 weeks regardless of responder status.
Arm/Group | Any AIN457 75 mg | Any AIN457 150 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 12/115 | 9/115 | 0/79
Other Adverse Events (participants affected / at risk) | 77/115 | 63/115 | 35/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=115) | Any AIN457 150 mg (N=115) | Placebo (N=79)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=115) | Any AIN457 150 mg (N=115) | Placebo (N=79)
Vertigo (Ear and labyrinth disorders) | 1 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 1
Dental caries (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 9 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 3 | 0
Nausea (Gastrointestinal disorders) | 4 | 6 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 6 | 1
Injection site pain (General disorders) | 5 | 1 | 1
Oedema peripheral (General disorders) | 1 | 4 | 2
Pyrexia (General disorders) | 5 | 0 | 0
Bronchitis (Infections and infestations) | 14 | 4 | 4
Cystitis (Infections and infestations) | 4 | 3 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 0
Influenza (Infections and infestations) | 5 | 2 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 25 | 23 | 8
Rhinitis (Infections and infestations) | 5 | 5 | 1
Sinusitis (Infections and infestations) | 2 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 9 | 3
Urinary tract infection (Infections and infestations) | 9 | 2 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 3 | 0
Weight increased (Investigations) | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 11 | 10 | 6
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Dizziness (Nervous system disorders) | 3 | 4 | 1
Headache (Nervous system disorders) | 6 | 10 | 2
Insomnia (Psychiatric disorders) | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 4 | 1
Hypertension (Vascular disorders) | 5 | 6 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to the decision (unrelated to safety) to discontinue the clinical development program for secukinumab in Rheumatoid Arthritis, with last patient last visit (LPLV) on 11-May-2015.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.